CLINICAL TRIAL: NCT00498095
Title: Experience of C4d Staining in Renal Allograft Biopsies
Brief Title: A Study on a New Staining Method (C4d Staining) of Transplanted Kidney Biopsies
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Other Study IDs: KW/EX/06-054; HARECCTR0500061
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Transplantation; Graft Rejection
Keywords: Delayed renal graft function; Acute renal allograft dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Renal biopsy

SUMMARY:
Patients who had received kidney transplantation may suffer from rejection. Recently, positive staining for C4d in kidney biopsies of malfunctioning transplant kidney is increasingly recognized as an important prognostic indicator of poorer long-term kidney outcome. Data is, however, lacking in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* All renal allograft biopsies performed in Princess Margaret Hospital (PMH) during the period 1st April 2003 to 31st August 2005 for unexplained acute renal dysfunction (Creatinine rise from baseline by ≥ 20%) or delayed graft function in the immediate post-transplantation period were included in the study. Both cadaveric and living-donor transplant allografts were included.

Exclusion Criteria:

* patients who were < 18 years' old at the time of renal biopsy or whose records were so incomplete that preclude meaningful analysis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All renal allograft biopsies performed in Princess Margaret Hospital from 1st April 2002 to 31st March 2006 on Chinese patients who were ≥ 18 years old were retrospectively reviewed. Renal transplantations were either cadaveric or living-donor related performed in Hong Kong or Mainland China. All recipients' sera produced negative cross-match tests with donor lymphocytes before transplantation and were ABO compatible. Finally, 52 renal biopsies were included. 38 (73.1%) of them were performed for unexplained acute renal deterioration whilst the rest were done for delayed graft function.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sze Kit Yuen, Dr, Principal Investigator — Department of Medicine & Geriatrics, ICU, Caritas Medical Centre
Locations (1):
- Princess Margaret Hospital, Hong Kong, China